CLINICAL TRIAL: NCT04601831
Title: A Phase I/II Trial of 'Re-Priming' Radiation Therapy for Relapsed/Refractory Non-Hodgkin Lymphoma Patients in Incomplete Response After Chimeric Antigen Receptor T-cell (CAR-T) Therapy
Brief Title: 'Re-Priming' RT After Incomplete Response to CAR-T in R/R NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kiran Kumar, Principal Investigator, Assistant Professor, Chief of Lymphoma & Pediatrics Radiation Oncology Service, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1106
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: CAR-T; Radiation therapy; NHL; DLBCL; RT
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Single-arm, open label, seamless phase I/II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation Therapy to all residual FDG-avid sites* (Experimental): All patients enrolled in the trial will receive focal radiation therapy (RT) to all* residual FDG-avid sites per Lugano criteria (Lugano 4-5) as noted on day 30 post-CAR-T PET/CT scan.
  *If >5 distinct sites, physician discretion will be allowed as to how many sites are treated, with recommendation that at least all symptomatic and bulky (>=7.5 cm in largest dimension) sites be treated.
  Interventions: Radiation: Focal radiation therapy (RT)

INTERVENTIONS:
Radiation: Focal radiation therapy (RT) — Radiation therapy for phase II:
  "Definitive" 40-50 Gy EQD2 (i.e. 30 Gy in 5 fractions)
  Hypofractionated regimen (i.e. 5 fractions in 1-2 weeks) recommended, but other fractionation schemes (10-20 fractions in 2-4 weeks) allowed.

SUMMARY:
This is a single-arm open-label phase I/II trial studying the safety and efficacy of focal 're-priming' radiation therapy (RT) to FDG-avid residual sites of disease in relapsed/refractory non-Hodgkin lymphoma (R/R NHL) patients with incomplete response (IR) to CAR T-cell therapy (CAR-T) by day 30 post-CAR-T PET/CT. We hypothesize that focal 're-priming' RT will be safe (phase I) and improve conversion to metabolic complete response (CR) by day 90 post-CAR-T PET/CT from 29% (historical control) to 58% (phase II).

DETAILED DESCRIPTION:
Early clinical trials of CAR-T in R/R NHL suggest that only ~40% of patients achieve CR by day 30 PET/CT evaluation. Of those who do not, the large majority (~70%) ultimately fail, while ~30% convert to CR after a median time of 64 days (range, 49-424). This group of patients, who have incomplete response on day 30 PET/CT after CAR-T and thus are most likely to fail CAR-T alone, may be the ideal target for early therapeutic intervention to 're-prime' CAR-T and convert them from IR to CR.

Preclinical and early clinical studies suggest potential immune augmentation when combining RT with CAR-T. Therefore, we propose a phase I/II clinical trial investigating the impact of RT to poor responding sites of disease after CD19-directed CAR-T in R/R NHL patients who are likely to fail CAR-T alone. We hypothesize that focal RT to residual FDG-avid sites of disease on day 30 PET/CT will improve the number of patients who convert to CR by day 90 PET/CT both through local cytotoxic effects as well as local and systemic synergistic effects through 're-priming' of CAR T-cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening
3. Biopsy-proven histological high-grade non-Hodgkin lymphoma, such as diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), or transformed follicular lymphoma.
4. Prior treatment with any CD19-directed CAR T-cell therapy, such as tisagenlecleucel (tisa-cel, Kymriah), axicabtagene ciloleucel (axi-cel, Yescarta), or lisocabtagene maraleucel (liso-cel).
5. Incomplete response noted on day 30 PET post-CAR-T, defined as not achieving CR per Lugano 2014 classification
6. Ability to understand and the willingness to sign a written informed consent
7. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

7.1 A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Prior "definitive" radiation therapy (40-50 Gy EQD2 with an α/β of 10) to one or more sites of incomplete response as noted on day 30 post-CAR-T PET/CT scan within the past one year. Prior "palliative" radiation therapy (<40 Gy EQD2) permissible at discretion of treating physician.
2. Intracranial site of incomplete response as noted on day 30 post-CAR-T PET/CT scan or any active central nervous system involvement by malignancy.
3. Active grade 3 or higher CRS or neurotoxicity related to CAR-T.
4. Patients with prior history of auto-immune disease or other contraindication to RT.
5. Patients with life expectancy < 3 months.
6. Psychiatric illness/social situations that would limit compliance with study requirements.
7. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events as Assessed by CTCAE v5.0, ASTCT Consensus Guidelines for CRS, and ASTCT ICANS Consensus Guidelines for Neurotoxicity [Phase 1: Safety and Tolerability] | 4 Months post CAR-T
  To determine the dose-limiting toxicity (DLT) and maximally tolerated dose (MTD) of RT to sites of incomplete response after CAR-T in patients with relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL).
  DLT rate will be defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade 4 or higher hematologic, grade 3 or higher dermatitis/burn, pneumonitis, enteritis, or other toxicity attributable to RT, as well as new grade 3 or higher cytokine release syndrome (CRS) per American Society for Transplantation and Cellular Therapy (ASTCT) consensus guidelines or grade 3 or higher neurotoxicity per ASTCT immune effector cell-associated neurotoxicity syndrome (ICANS) consensus guidelines for adults. For those who had prior stem cell transplant (SCT), DLT will also be defined by grade C or D graft-versus-host-disease (GVHD) per International Bone Marrow Transplant Registry (IBMTR) grading system.
Rate of Metabolic Complete Response (CR) on Day 90 Post-CAR-T PET/CT scan per Lugano 2014 Classification [Phase 2: Efficacy] | Day 90 post CAR-T
  To assess the efficacy of adding RT to sites of incomplete response after CAR-T in R/R NHL patients by determining the rate of metabolic complete response (CR) at day 90 post-CAR-T PET/CT scan, assessed per Lugano 2014 classification.

SECONDARY OUTCOMES:
Response rates of individual sites | Day 90 PET post-CAR-T
  To determine the rates of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), and overall response rate (ORR) of all irradiated and un-irradiated sites on day 90 PET post-CAR-T.
Duration of response (DOR) in Participants with Any Response as Noted on Day 90 Post-CAR-T PET/CT | 1 year
  To determine the duration of response (DOR) for patients who have any response as noted on day 90 PET post-CAR-T, defined as time from day 90 post-CAR-T PET/CT to first PET/CT scan showing progression.
Progression free survival (PFS) | 1 year
  To determine the progression free survival (PFS) for all patients at 1-year post-CAR-T
Overall survival (OS) | 1 year
  To determine the overall survival (OS) for all patients all patients at 1-year post-CAR-T

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Kumar, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States